CLINICAL TRIAL: NCT05820581
Title: Characterization of Mentalization Profiles Related to Emotional Regulation Among Teenagers With Behavioral Disorders
Acronym: CARMEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/646
Record Dates: First submitted 2023-03-27; First posted 2023-04-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Adolescent Behavior Disorder; Eye Movements
Keywords: Mentalisation; Emotion regulation; Adolescents; Neurophysiological parameters
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mentalisation (Experimental): 4 mentalisation groups will be defined: hypomentalisation, hypermentalisation, mentalisation correct and lack of mentalisation
  Interventions: Behavioral: Mentalisation

INTERVENTIONS:
Behavioral: Mentalisation — Hypomentalisation, hypermentalisation, correct mentalisation, lack of mentalisation

SUMMARY:
Behavioral disorders in adolescents are defined by a set of diverse behaviors (such as aggressiveness, agitation, clastic crisis, running away and endangerment) whose common characteristic is the predominance of action/ mentalization. These disorders are associated with significant morbidity and high mortality linked to a high rate of suicide or attempted suicide. Behavioral disorders are also associated with an alteration of mentalizing capacities, that is the psychic process by which the adolescent imagines and interprets his behavior and that of others on the basis of mental states such as needs, desires, beliefs or feelings. The disorders are also associated with emotional dysregulation. To date, the psychopathological processes underlying behavioral disorders in adolescents are unknown and prevent from offering appropriate psychological care. Thus, it seems essential to characterize this clinical population by integrating both its intrapsychic representations and the physiological parameters of emotional regulation associated with it.

This project is a first step towards a larger-scale research project aimed at evaluating treatment by TBM (therapies based on mentalization) in adolescents with behavioral disorders.

DETAILED DESCRIPTION:
Behavioral disorders in adolescents are defined by a set of behaviors (such as aggressiveness, agitation, clastic crisis, running away and endangerment) whose common characteristic is the predominance of action over mentalization and opposition to normal socialization processes.

These disorders are associated with significant morbidity and high mortality linked to a high rate suicide or attempted suicide. Behavioral disorders in adolescence are linked to defects of mentalization (i.e. the psychic process by which the adolescent imagines and interprets his behaviors and to alterations in emotional regulation capacities. This emotional dysregulation has several components, including motor and physiological components. Moreover, this dysregulation is constructed in a dynamic process linked to the environment, including the adolescent's relationship with parents. To date, the psychopathological processes underlying behavioral disorders in the teenager are unknown, which prevents from offering appropriate psychological care. Thus, it seems essential to characterize adolescents behavior, by integrating both mentalizing capacities, the physiological parameters of their emotional regulation and the interactive patterns with their parents. This approach allow to overcome the difficulty of adolescents to use words to express what they feel and thus to understand their psychic functioning and the strategies, which they put in place to regulate their emotions.

This study is a monocentric cross-sectional descriptive observational study.

Objectives of this study is to describe the mentalization profiles of adolescents with mental disorders behavior and to evaluate:

* Oculomotor parameters of emotional regulation
* Physiological parameters of emotional regulation (Electrodermal Activity, RED)
* Self-assessed mentalizing abilities (RFQ-Y scale)
* Emotional regulation (DERS scale)
* The emotional and behavioral functioning of adolescents (YSR scale)
* Attachment characteristics of adolescents (ARSQ scale)
* The interactions of the adolescent with his parent (GPACS scale)
* Parental reflexive capacities (RFQ scale). This research was developed to support a comprehensive understanding of adolescent processes with the integration of bio-neuro-social parameters.

The aim of this study is to establish mentalization profiles of the clinical population of adolescents with behavioral disorders and their neurophysiological correlates of emotional regulation.

These first data are essential for a better understanding of this clinical population and a starting point for future research; particularly to develop therapies based on mentalization in this population and to evaluate their effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Teenage girls or boys aged 12 to 17
* Adolescent(s) with externalized behavioral disorder(s):

running away, suicide attempts, self-aggression (scarification, self-mutilation), taking drugs, hetero-aggressive behavior, theft, conduct disorders sexual, oppositional behavior, lies, clastic anger.

* Non-objection of the adolescent to participate in the study.
* Written consent of the two holders of parental authority

Exclusion Criteria:

* Intellectually disabled
* Autism Spectrum Disorder
* Psychotic disorder

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
eye fixation duration evaluated with eyes tracker | 12 months
  fixation duration (time in millisecond)
eye dwell time evaluated with eyes tracker | 12 months
  dwell time (time in millisecond)
eye fixation count evaluated with eyes tracker | 12 months
  fixation count ( time in millisecond)

SECONDARY OUTCOMES:
MASC Score | 12 months
  Mentalization score
YSR score | 12 months
  youth self report score
RFQ-Y score | 12 months
  Reflective Function Questionnaire for Youth
DERS score | 12 months
  Difficulties in Emotion Regulation Scale (DERS)
ARSQ score | 12 months
  Adolescent relationship scale questionnaire
parent's RFQ score | 12 months
  Reflective Functioning Questionnaire for parents
GPACS interaction evaluation | 12 months
  General Practitioner Attitudes and Confidence Scale is a tool to measure confidence and attitude.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Pozet, MS, Study Chair — CHU Besancon, DRCI
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szymanska M, Monnin J, Tio G, Vidal C, Girard F, Galdon L, Smith CC, Bifulco A, Nezelof S, Vulliez-Coady L. How do adolescents regulate distress according to attachment style? A combined eye-tracking and neurophysiological approach. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Mar 8;89:39-47. doi: 10.1016/j.pnpbp.2018.08.019. Epub 2018 Aug 27. PMID 30165119
- [Background] Taubner S, Volkert J, Gablonski TC, Rossouw T. [Mentalization-Based Treatment for Adolescents with Borderline Personality Disorder - Concept and Efficacy]. Prax Kinderpsychol Kinderpsychiatr. 2017 Jul;66(6):423-434. doi: 10.13109/prkk.2017.66.6.423. German. PMID 28701091
- [Background] Sharp C, Pane H, Ha C, Venta A, Patel AB, Sturek J, Fonagy P. Theory of mind and emotion regulation difficulties in adolescents with borderline traits. J Am Acad Child Adolesc Psychiatry. 2011 Jun;50(6):563-573.e1. doi: 10.1016/j.jaac.2011.01.017. Epub 2011 Mar 9. PMID 21621140
- [Background] Sharp C, Ha C, Carbone C, Kim S, Perry K, Williams L, Fonagy P. Hypermentalizing in adolescent inpatients: treatment effects and association with borderline traits. J Pers Disord. 2013 Feb;27(1):3-18. doi: 10.1521/pedi.2013.27.1.3. PMID 23342954
- [Background] Quek J, Bennett C, Melvin GA, Saeedi N, Gordon MS, Newman LK. An investigation of the mentalization-based model of borderline pathology in adolescents. Compr Psychiatry. 2018 Jul;84:87-94. doi: 10.1016/j.comppsych.2018.04.005. Epub 2018 Apr 14. PMID 29727808